CLINICAL TRIAL: NCT02425683
Title: A Randomized, Phase II Study of High-Risk Colorectal Cancer Patients (Stage IIIC) Treated With Either Regorafenib or Standard of Care (No Treatment) After Adjuvant FOLFOX
Brief Title: Study of Colorectal Cancer Patients (Stage IIIC) With Either Regorafenib or Standard of Care (No Treatment) After Adjuvant FOLFOX
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: insufficient accrual
Sponsor: US Oncology Research (Industry)
Collaborators: Bayer Healthcare Pharmaceuticals, Inc./Bayer Schering Pharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 13050
Record Dates: First submitted 2015-04-21; First posted 2015-04-24 (Estimated); Last update posted 2020-02-10 (Actual); Status verified 2020-02

CONDITIONS: Colorectal Neoplasms; Adenocarcinoma of the Colon; Adenocarcinoma of the Rectum
Keywords: Colon Cancer; Rectal Cancer; Colorectal Cancer; Stage IIIC Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms; Colonic Neoplasms; Rectal Neoplasms | interventions — regorafenib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Regorafenib (Experimental): Regorafenib 120 or 160 mg by mouth every day for the first 21 days of each 28-day cycle. If the dose is tolerated during the first 2 cycles in the 120 mg group, in Cycle 3 the 120 mg dose will be increased to 160 mg by mouth each day for the first 21 days of each 28-day cycle for 4 more cycles for a total of 6 cycles or 6 months of therapy.
  Interventions: Drug: Regorafenib
- Standard of Care (No Treatment) (No Intervention): No study drug (which is the standard care for Stage IIIC colorectal cancer patients after they've received FOLFOX chemotherapy).

INTERVENTIONS:
Drug: Regorafenib — 120 mg or 160 mg by mouth each day for first 21 days of each 28-day cycle, for maximum of 6 cycles
  Other Names: Stivarga; BAY 73-4506
  Arms: Regorafenib

SUMMARY:
This study, for patients who have Stage IIIC colorectal cancer and who underwent 5-fluorouracil/leucovorin with oxaliplatin (FOLFOX) chemotherapy after surgery, will test to see if regorafenib given after the completion of FOLFOX improves treatment, compared to standard of care (SOC), which is no further treatment.

DETAILED DESCRIPTION:
Patients with Stage IIIC colon cancer have a 5-year survival rate of 28%. Stage III colon cancer indicates that lymph nodes are involved.

Adjuvant FOLFOX only reduces the risk of recurrence of colorectal cancer by 40%, so almost 50% of patients still die from the disease. It is estimated that 50% of the patients relapse within 18 months.

Because the prognosis of colorectal cancer is dependent on disease stage and because metastatic disease is incurable, the concept of adding regorafenib to adjuvant FOLFOX has been developed to allow patients with high-risk colorectal cancer the best chance of cure.

It is proposed to treat high-risk colorectal patients (Stage IIIC [T4a, N2a, M0] or [T3-4a,N2b, M0], or [T4b, N1-N2, M0] per American Joint Committee on Cancer [AJCC] 7th ed.) selected from the iKnowMed (iKM) electronic health records database who have completed adjuvant FOLFOX. This feasibility study is to find the starting dose of regorafenib and estimates that at least 75% of the patients will be able to tolerate the full dose of regorafenib after receiving adjuvant FOLFOX.

Patients will be randomly assigned to regorafenib or to SOC (no treatment). In order to test the best tolerated starting dose, the first 50 patients will receive regorafenib and will be randomized 1:1 to either 120 mg by mouth (PO) or 160 mg PO. If the 120 mg dose is well tolerated and the toxicities are not severe (Grade 2 or less) upon the completion of cycle 2, the dose will be increased to 160 mg starting with Cycle 3. Registration and randomization of patients will resume after the 26th then after the 50th patient completes 3 cycles of study treatment. The Data Safety Monitoring Board (DSMB) will meet after the 26th patient completes 3 cycles of treatment and the second meeting will take place after the 50th patient completes 3 cycles. If needed, a third DSMB meeting will be scheduled. The remaining 214 patients will be randomized 2:3 to the decided starting dose versus SOC.

In addition, evaluating the Texture (spatial variations in pixel intensity) in computed tomography (CT) scans might help predict the risk of recurrence. Therefore, CT disks will be sent to Imaging Endpoints Core Lab, Scottsdale, AZ, where the TexRAD platform (a software algorithm) will be used for analysis.

ELIGIBILITY:
Inclusion Criteria:

* A signed Patient Authorization Form (HIPAA) has been obtained prior to registration
* Subjects must be able to understand and be willing to sign the written informed consent form. A signed informed consent form must be appropriately obtained prior to the conduct of any trial-specific procedure.
* Age ≥ 18 years.
* Stage IIIC colorectal cancer (T4a, N2a, M0) or (T3-4a, N2b, M0), or (T4b, N1- N2, M0) (per AJCC 7th ed).
* Must have started adjuvant FOLFOX chemotherapy within 8 weeks of resection for colorectal carcinoma
* CT scan that demonstrates no evidence of disease (NED) after completion of adjuvant therapy Note: This CT scan will also be used for Texture analysis.
* Received FOLFOX within 6 weeks before starting regorafenib
* Eastern Cooperative Oncology Group (ECOG) performance status 0-1
* Life expectancy of at least 12 weeks (3 months).
* Complete Metabolic Profile (CMP) within normal limits
* Adequate bone marrow, liver, and renal function as assessed by the following laboratory requirements:

  * Total bilirubin ≤ 1.5 x the upper limits of normal (ULN)
  * Alanine aminotransferase (ALT) and aspartate amino-transferase (AST) ≤ 2.5 x ULN
  * Alkaline phosphatase limit ≤ 2.5 x ULN
  * Lipase ≤ 1.5 x ULN
  * Serum creatinine ≤ 1.5 x ULN
  * International normalized ratio (INR)/ Partial thromboplastin time (PTT) ≤ 1.5 x ULN. (Subjects who are prophylactically treated with an agent such as warfarin or heparin will be allowed to participate provided that no prior evidence of underlying abnormality in coagulation parameters exists. Close monitoring of at least weekly evaluations will be performed until INR/PTT is stable based on a measurement that is pre-dose as defined by the local standard of care.
  * Platelet count ≥ 100,000 /mm3, hemoglobin (Hb) ≥ 9 g/dL, absolute neutrophil count (ANC) ≥ 1500/mm3. Blood transfusion to meet the inclusion criteria will not be allowed.
* Normal carcinoembryonic antigen (CEA) prior to study entry
* Glomerular filtration rate (GFR) ≥ 60 mL/min/1.73 m2 according to the Modified Diet in Renal Disease (MDRD) abbreviated formula.
* Women of childbearing potential must have a negative serum pregnancy test performed within 7 days prior to the start of study drug. Post-menopausal women (defined as no menses for at least 1 year) and surgically sterilized women are not required to undergo a pregnancy test. The definition of adequate contraception will be based on the judgment of the investigator.
* Subjects (men and women) of childbearing potential must agree to use adequate contraception beginning at the signing of the informed consent form (ICF) until at least 3 months after the last dose of study drug. The definition of adequate contraception will be based on the judgment of the principal investigator or a designated associate.
* Subject must be able to swallow and retain oral medication.
* Discretionary use of growth factors allowed

Exclusion Criteria:

* Previous assignment to treatment during this study. Subjects permanently withdrawn from study participation will not be allowed to re-enter study.
* Uncontrolled hypertension (systolic pressure >140 mm Hg or diastolic pressure > 90 mm Hg [NCI-Common Toxicity Criteria for Adverse Effects (CTCAE) v4.03] on repeated measurement) despite optimal medical management.
* Evidence of remaining tumor
* Has local or distant metastasis
* Previous antiangiogenic treatment
* Abnormal hematological, renal, or liver function
* Impaired pulmonary function
* Evidence of ≥ Grade 2 neuropathy
* Active or clinically significant cardiac disease including:

  * Congestive heart failure - New York Heart Association (NYHA) > Class II.
  * Active coronary artery disease.
  * Cardiac arrhythmias requiring anti-arrhythmic therapy other than beta blockers or digoxin.
  * Unstable angina (anginal symptoms at rest), new-onset angina within 3 months before randomization, or myocardial infarction within 6 months before randomization.
* Evidence or history of bleeding diathesis or coagulopathy.
* Any hemorrhage or bleeding event ≥ NCI CTCAE Grade 3 within 4 weeks prior to start of study medication.
* Subjects with thrombotic, embolic, venous, or arterial events, such as cerebrovascular accident (including transient ischemic attacks), deep vein thrombosis, or pulmonary embolism within 6 months of start of study treatment.
* Subjects with any previously untreated or concurrent cancer that is distinct in primary site or histology from breast cancer except cervical cancer in-situ, treated basal cell carcinoma, or superficial bladder tumor. Subjects surviving a cancer that was curatively treated and without evidence of disease for more than 3 years before randomization are allowed. All cancer treatments must be completed at least 3 years prior to study entry (ie, signature date of the informed consent form).
* Patients with phaeochromocytoma.
* Known history of human immunodeficiency virus (HIV) infection or current chronic or active hepatitis B or C infection requiring treatment with antiviral therapy.
* Ongoing infection > Grade 2 NCI-CTCAE v4.03.
* Presence of a non-healing wound, non-healing ulcer, or bone fracture.
* Dehydration Grade ≥ 1 NCI-CTCAE v4.03.
* Patients with seizure disorder requiring medication.
* Persistent proteinuria ≥ Grade 3 NCI-CTCAE v4.03 (> 3.5 g/24 hrs, measured by urine protein: creatinine ratio on a random urine sample).
* Interstitial lung disease with ongoing signs and symptoms at the time of informed consent.
* Pleural effusion or ascites that causes respiratory compromise (≥ NCI-CTCAE version 4.03 Grade 2 dyspnea).
* History of organ allograft (including corneal transplant).
* Known or suspected allergy or hypersensitivity to any of the study drugs, study drug classes, or excipients of the formulations given during the course of this trial.
* Any malabsorption condition.
* Women who are pregnant or breast-feeding.
* Any condition which, in the investigator's opinion, makes the subject unsuitable for trial participation.
* Substance abuse, medical, psychological or social conditions that may interfere with the subject's participation in the study or evaluation of the study results.
* Concurrent anti-cancer therapy (chemotherapy, radiation therapy, surgery, immunotherapy, biologic therapy, or tumor embolization) other than study treatment (regorafenib, other agents being investigated in combination with regorafenib).
* Prior use of regorafenib.
* Concurrent use of another investigational drug or device therapy (ie, outside of study treatment) during, or within 4 weeks of trial entry (signing of the informed consent form).
* Major surgical procedure, open biopsy, or significant traumatic injury within 28 days before start of study medication.
* Therapeutic anticoagulation with Vitamin-K antagonists (eg, warfarin) or with heparins and heparinoids.

  o However, prophylactic anticoagulation as described below is allowed:
  * Low dose warfarin (1 mg orally, once daily) with PT-INR ≤ 1.5 x ULN is permitted. Infrequent bleeding or elevations in PT-INR have been reported in some subjects taking warfarin while on regorafenib therapy. Therefore, subjects taking concomitant warfarin should be monitored regularly for changes in PT, PT-INR, or clinical bleeding episodes.
  * Low dose aspirin (≤ 100 mg daily).
  * Prophylactic doses of heparin.
* Use of any herbal remedy (eg, St. John's wort [Hypericum perforatum]) Note: Granulocyte colony-stimulating factor (G-CSF) and other hematopoietic growth factors may be used in the management of acute toxicity, such as febrile neutropenia, when clinically indicated or at the investigator's discretion. However, they may not be substituted for a required dose reduction. Subjects are permitted to take chronic erythropoietin.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2015-03-26 (Actual); Primary Completion 2017-09-21 (Actual); Study Completion 2017-09-21 (Actual)

PRIMARY OUTCOMES:
Starting Dose of Regorafenib | 1 year
  To find the starting dose of regorafenib. The first 50 patients will be randomly assigned to receive regorafenib either 120 mg or 160 mg by mouth daily for 1st 21 days of each 28-day cycle for two cycles. Based on safety profile review of adverse events, a final starting dose will be selected for remaining patients assigned to regorafenib.
Number of Patients Completing Full 6 Cycles | 4.5 years
  To have at least 75% of enrolled Stage IIIC high-risk colorectal cancer patients in each treatment arm complete the full duration of adjuvant therapy.

SECONDARY OUTCOMES:
Overall survival | 4.5 years
  To estimate overall survival (OS) in each treatment arm
Number of Adverse Events (AEs) | 4.5 years
  To estimate Adverse Events (AE) in each treatment arm.
Disease-free survival (DFS) | 4.5 years
  To determine the association between Texture results in CT scans and DFS in a retrospective subanalysis.

CONTACTS AND LOCATIONS:
Overall Officials: Thomas H. Cartwright, MD, Principal Investigator — US Oncology Research, McKesson Specialty Health
Locations (1):
- 24 Sites, Including Dallas, TX, Ocala, FL, Denver, CO, Florida, United States